CLINICAL TRIAL: NCT03473587
Title: Promoting Colorectal Cancer Screening in Rural Emergency Departments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Kentucky (Other)
Responsible Party: Principal Investigator, Jennifer Hatcher, Principal Investigator, University of Kentucky
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MCC-14-0681-P1H
Record Dates: First submitted 2018-01-18; First posted 2018-03-22 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Motivational Interviewing; Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interview (Experimental): Subjects will engage in a brief motivational interview to establish an action plan and discuss follow-up interviews a 3 and 6 months post ED visit
  Interventions: Behavioral: Motivational interview
- Standard of Care (Active Comparator): Subjects will be provided a standard of care colorectal cancer screening brochure at the time of ED visit
  Interventions: Behavioral: Standard of care

INTERVENTIONS:
Behavioral: Motivational interview — A lay health advisor will engage the subject in a motivational interview to promote the importance of colorectal cancer screening
  Arms: Motivational Interview
Behavioral: Standard of care — A lay health advisor will provide the subject with a brochure promoting the importance of colorectal cancer screening
  Arms: Standard of Care

SUMMARY:
This trial will compare the effects of a culturally targeted intervention designed to assist participants to identify and overcome individual barriers to colorectal cancer (CRC) and to promote CRC screenings using motivational interviewing (Ml) delivered by a lay health advisor (LHA) compared to the current standard-of-care (distribution of a brochure describing CRC screening services offered by the hospital) on CRC screening compliance.

DETAILED DESCRIPTION:
The specific aim of this project is to adapt and pilot a tailored intervention to promote CRC screenings in a rural Appalachian Kentucky emergency department (ED) in order to: (a) evaluate the feasibility of providing a cancer screening promotion intervention in an emergency department (ED) that serves a rural Appalachian community; and (b) assess the effects of the intervention on barriers to CRC screening, stage of readiness to screen and CRC screening engagement. The first phase of the project will involve the adaptation and pretesting of the intervention. This phase will take approximately 6 months. The second phase of the project will involve piloting the intervention and evaluating its efficacy and feasibility and will take place over the following 18 months. We will conduct a randomized controlled trial to examine the efficacy and feasibility of delivering the LHA delivered MI intervention to promote CRC screening in persons waiting in a rural Appalachian emergency department (ED) for non urgent complaints. We will evaluate efficacy by measurement of CRC screening status at baseline and three and six months post intervention.

ELIGIBILITY:
Inclusion Criteria:

1. 50+ years of age
2. Rural Appalachian resident
3. No personal history of colorectal cancer
4. No cognitive impairment
5. Ability to speak and understand English
6. Has not had one of the following colorectal cancer screening tests--

   1. Fecal Occult Blood Test within the past year
   2. Flexible sigmoidoscopy within the past five years, or
   3. Colonoscopy within the past ten years

Exclusion Criteria:

-

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 191 (Estimated)
Dates: Start 2014-11-07 (Actual); Primary Completion 2018-05-30 (Estimated); Study Completion 2018-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in colorectal cancer screening rate | 6 months
  Number of participants that seek out colorectal cancer screening after a motivational interview with a lay health advisor compared to standard of care (being provided a screening brochure)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Hatcher, RN, PhD, Principal Investigator — University of Kentucky
Locations (1):
- St. Clair Regional Medical Center, Morehead, Kentucky, United States